CLINICAL TRIAL: NCT07046598
Title: Is The Level of Muscle Damage After The Drop Jump Protocol Affected By Body Weight and BMI?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Melike Nur Eroğlu (Other)
Responsible Party: Sponsor-Investigator, Melike Nur Eroğlu, Lecturer, Sakarya Applied Sciences University
Organization: Sakarya Applied Sciences University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SakaryaAppliedSciencesU
Record Dates: First submitted 2025-06-14; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Body Mass Index; Physical Exertion; Muscle Damage; Creatine Kinase; Lactate Dehydrogenases
Keywords: drop jump; muscle damage; creatine kinase; lactate dehydrogenase; body mass index; plyometric exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal Weight Group (Experimental): Participants with a Body Mass Index (BMI) between 18 and 24 kg/m². Subjects in this group performed a standardized drop jump (DJ) protocol consisting of 100 total jumps from a 60 cm platform. Muscle damage markers (Creatine Kinase and Lactate Dehydrogenase) were measured pre-exercise, immediately post-exercise, and 24 hours post-exercise.
  Interventions: Behavioral: Drop Jump Protocol
- Overweight Group (Experimental): Participants with a Body Mass Index (BMI) between 25 and 35 kg/m². Subjects in this group performed the same standardized drop jump (DJ) protocol as the normal weight group. Blood samples were collected at three time points to evaluate changes in muscle damage markers (Creatine Kinase and Lactate Dehydrogenase).
  Interventions: Behavioral: Drop Jump Protocol

INTERVENTIONS:
Behavioral: Drop Jump Protocol — A standardized drop jump (DJ) protocol involving 100 total jumps from a 60 cm platform. Participants performed five sets of 20 jumps, with a 10-second rest between jumps and a 2-minute rest between sets. The protocol was designed to induce muscle damage through eccentric loading.

SUMMARY:
This study investigated whether muscle damage induced by a drop jump protocol varies based on participants' body weight and BMI. Fifty healthy adults were divided into normal-weight and overweight groups. All participants completed a standardized drop jump protocol, and blood samples were collected before, immediately after, and 24 hours after exercise. Creatine kinase (CK) and lactate dehydrogenase (LDH) levels were analyzed as biomarkers of muscle damage.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18-30
* Normal or overweight BMI (18-35 kg/m²)
* At least 2 days/week of physical activity
* No regular jump training

Exclusion Criteria:

* Use of medications or supplements
* History of musculoskeletal injury
* Smoking or alcohol consumption during study period

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2024-11-08 (Actual); Study Completion 2024-11-22 (Actual)

PRIMARY OUTCOMES:
Change in Creatine Kinase (CK) Levels | Baseline (pre-exercise), immediately post-exercise, and 24 hours post-exercise
  Serum creatine kinase (CK) concentrations measured at three time points: before the exercise protocol, immediately after the protocol, and 24 hours post-exercise. CK is a biomarker of muscle damage. Blood samples were analyzed using a standard biochemical analyzer.
Change in Lactate Dehydrogenase (LDH) Levels | Baseline (pre-exercise), immediately post-exercise, and 24 hours post-exercise
  Serum lactate dehydrogenase (LDH) concentrations measured at three time points: before the exercise protocol, immediately after the protocol, and 24 hours post-exercise. LDH is used to evaluate exercise-induced muscle damage. Blood samples were centrifuged and analyzed using standardized laboratory techniques.

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya University of Applied Sciences, Faculty of Sport Sciences, Exercise and Sports Sciences Education, Application and Research Centre, Serdivan, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yeniyol B, Pancar S, Soylu Y, Birinci YZ, Eroglu MN, Fernandez-Elias VE. The overlooked risk in drop jump protocols: higher body weight as a catalyst for increased muscle damage. BMC Sports Sci Med Rehabil. 2025 Sep 29;17(1):278. doi: 10.1186/s13102-025-01330-z. PMID 41024229

DOCUMENTS (1):
  • Informed Consent Form (2024-10-15): https://cdn.clinicaltrials.gov/large-docs/98/NCT07046598/ICF_000.pdf